CLINICAL TRIAL: NCT02873559
Title: Effect of PROGRESSive Resistance Training, Protein Supplements and Testosterone in Older Frail Men With Testosterone Deficiency (PROGRESS Trial)
Brief Title: Effect of PROGRESSive Training and Teststerone in Older Frail Men
Acronym: PROGRESS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Rune Skovgaard Rasmussen, Neuropychologist, Ph.D., associate professor, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ethical protocol H-16020521
Record Dates: First submitted 2016-08-12; First posted 2016-08-19 (Estimated); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Muscle Weakness
Keywords: older; frail; men; progressive muscle training; muscle training; exercise; testosterone
MeSH Terms: conditions — Muscle Weakness; Multiple Endocrine Neoplasia Type 1; Motor Activity | interventions — Testosterone; Autogenic Training

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Controls (No Intervention): A control group, which is 20 weeks with placebo injections without training.
- Testosterone (Experimental): A testosterone group given 20 weeks on testosterone injections without training
  Interventions: Drug: testosterone
- Training (Experimental): A Training Group, which is 20 weeks with placebo injections and 16 weeks of progressive resistance training supplemented with vitamin D and protein supplements
  Interventions: Other: Progressive muscle training
- Testosterone and training (Experimental): A combination group that is 20 weeks with testosterone injections and 16 weeks of progressive resistance training supplemented with vitamin D and protein supplements
  Interventions: Drug: testosterone; Other: Progressive muscle training

INTERVENTIONS:
Drug: testosterone — Testosterone supplemented in 5 months
  Arms: Testosterone; Testosterone and training
Other: Progressive muscle training — Progressive muscle training during 4 months
  Other Names: Training
  Arms: Testosterone and training; Training

SUMMARY:
In this scientific clinical investigation we will test whether testosterone and progressive resistance training can improve muscle strength and reduce the risk of falls in older men. In addition, we will examine whether this treatment improves quality of life, functional capacity, including sexual function and counteracts depression. Such a project have not been performed earlier.

DETAILED DESCRIPTION:
Project background: In Denmark more than 1,000 people each year die of a fall, which is more than five times as many dying in traffic accidents. Fall accidents are also the leading cause of traumatic brain injury and is a relatively unnoticed problem, although this type of accidents causes more hospital bed days than all other accidents combined.

Annually, almost half of the 375,000 elderly Danes over 75 years of age and relatively three times as many of the approximately 40,000 elderly people in nursing homes fall every year, causing over 40,000 hospital contacts annually. Ten percent of all elderly people hospitalized each year because of a fall, mostly with fractures, for which the risk increases fivefold after a fall. In Denmark there are now now around 1 million people over 65 years of age. Over the next 25 years we will experience a 50% growth to 1.5 million people over 65 years of age.

Injury, disability and death caused by falls is therefore a widespread and growing human and societal problem. Many will never recover completely and will therefore need help to cope with everyday life. After the first fall risk increase for repeated falls. Especially for older people living in their own homes permanent or temporary disabilities results in a severe deterioration of the quality of life. Treatment of falls is also a significant financial burden on health and social care.

The main reason for the decline is muscle weakness. Muscle weakness leads to greatly increased risk of falling, decreased quality of life and functional capacity. Musclemass and -power decrease about 40 percent from age 20 to 80 years old.

Recent studies have shown that even 90-year-old persons can double their muscle strength by intensive training just three times per week. The level of the male sex hormone testosterone decreases with age and leads to impaired muscle mass. Twenty percent of men over 60 and 50 percent over 80 years, a low level of testosterone in total equivalent to more than 100,000 Danes. From the human and socio-economic perspective, it is important to find treatments that can enhance function in the elderly.

ELIGIBILITY:
Inclusion Criteria:

Living in their own home or in sheltered accommodation. Independent gait possible. with tool. Capable of stand-up and sit in a chair at least 8 times in 30 sec. There must be at least 3 symptoms or objective findings of low testosterone . Serum testosterone <10nmol /L as the average of two independent measurements

-

Exclusion Criteria:

Known or previous prostate cancer. Abnormally elevated serum PSA (PSA = prostate specific antigen) corresponding to PSA> 5 ng / ml or PSA> 0.15 ng / ml / cc (relative to the prostatic volume in cubic centimeters (cc)). Hæmatomacrose. Heart disease in the form of: peri-, myo-, or endocarditis, angina, severe heart failure (NYHA class III and IV), severe hypertension (systolic blood pressure> 180 or diastolic BT> 105 mmHg after antihypertensive therapy). Dyspnoea at rest. Liver (AST> 2 x ULN) or renal impairment (serum creatinine> 200 micromoles / L). Severe and insufficiently treated epilepsy or migraine. Insulin treatment. Previous or current bifosfonat-, fluoride, HRT, SERM-, strontium, teraparatid- or more than 3 weeks of prednisolone. Joint disease with acute inflammation. Active cancer disease in chemo- or radiotherapy. Bone metabolic disease apart from age-related osteoporosis. Autoimmune diseases, chronic systemic diseases (cirrhosis, AIDS, chronic renal failure). Primary testosterone deficiency in the form of testicular dysgenesis, Klinefelter syndrome (47, XXY), 46, XX males, LH-resistance, the Y chromosome deletions, other sex chromosome abnormalities ,. Significant abuse, mental illness, dementia, physical disability with inability to implement intervention or tests or to give informed consent. Contraindications to testosterone undecanoate is included in the exclusion criteria, such as. presence of liver tumors, breast and prostate cancer, as subjects will be examined before the trial starts.

Min Age: 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 192 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2023-03 (Actual)

PRIMARY OUTCOMES:
Stand-up-and Sit-test | up to 5 months (at study completion)
  It is a measure of overall strength in the lower extremities. Result of the test is defined as the number of times the participant can stand up and sit from a chair in 30 seconds. There is a good correlation (r = 0.78) with a leg press and an acceptable test-retest reliability (ICC = 0.86).

SECONDARY OUTCOMES:
Frequency and severity of falls via questionaire | At baseline, 1 month, 5 months (at study completion)
  included in the monitoring of adverse events.
Balance ability, | At baseline, 1 month, 5 months (at study completion)
  Tandem Test containing three starting positions: 1) Standing with feet together, standing in the semi-tandem position and standing in the tandem stand. coupled with decrease risk of fall.
Avlund mobility scale | At baseline, 1 month, 5 months (at study completion)
  Questions about experiencing fatigue and support needs of ordinary everyday activities. Avlund mobility scale is correlated with the isometric muscle strength, simple function tests , increased risk of hospitalization and mortality
Leg extensor Power Rig test | At baseline, 1 month, 5 months (at study completion)
  An instrument for measuring muscle strength in the lower extremities.
Isometric muscle strength | At baseline, 1 month, 5 months (at study completion)
  Measurement of isometric muscle strength m. quadriceps in a seated leg press.
Armflexion Test: | At baseline, 1 month, 5 months (at study completion)
  Measures of overall strength in the upper extremities. The number of times the participant can inflect the elbow with dumbbell is measured in 30 sec.
2-minute knee lift test: | At baseline, 1 month, 5 months (at study completion)
  Measures aerobic capacity in the elderly. Number of high knee lifts in 2 minutes.
2,45minute up-and-go test: | At baseline, 1 month, 5 months (at study completion)
  Target for basic mobility in the elderly. Time it takes to rise from a chair, walk around a cone 2,45m away, go back and sit down again. Moderate to good correlation between the corresponding 3m test and Berg Balance Scale (r = 0.81), walking speed (r = 0.61) and Barthel index (r = 0.78) and a good test-retest- reliability (ICC = 0.98).
DXA scan | At baseline, 1 month, 5 months (at study completion)
  Lean body mass. Measurement of fat and fat-free mass and total bone mass (BMC). Executed only at baseline and at study end.
Bone Mineral Density | At baseline, 1 month, 5 months (at study completion
  Of the spine, distal forearm bilaterally, total hip bilaterally and in the skeleton as a whole (total body). In case of osteoporosis treatment will be initiated following the department's usual guidelines, which can blur the results for bone density.
Major Depression Inventory (MDI): | At baseline, 1 month, 5 months (at study completion)
  Questionnaire on depression and mental well-being.
Montreal Cognitive Assessment (MoCA): | At baseline, 1 month, 5 months (at study completion)
  A cognitive screening test that provides an estimate of the intellectual functioning; This test is also sensitive to mild cognitive problems and dementia.
Quality of Life EQ-5D: | At baseline, 1 month, 5 months (at study completion)
  Questionnaire on the experienced quality of life.
Modified PISQ-12: | At baseline, 1 month, 5 months (at study completion)
  An assessment of sexual performance (potency) and sexual desire. There are previously found improved sexual function, mood, muscle strength and body composiAn evaluation questionnaire of sexual function
Aastrands Test: | At baseline, 1 month, 5 months (at study completion)
  Sub-maximal fitness test performed on a treadmill. Includes monitoring heart rate
Measurements of the Heart Rate Variability (HRV) | At baseline, 1 month, 5 months (at study completion)
  Studies have indicated that hypogonodal men can improve the Heart Rate Variability by testosterone treatment
Dual-energy X-ray absorptiometry | At baseline, 1 month, 5 months (at study completion)
  Measurement of the body composition bioimpedance.
Safety parameters - blood pressure | Measured every four weeks through the study (for 5 months)
  Blood pressure. Blood samples: Serum testosterone, hemoglobin, hematocrit, lipid profile, Potassium, Natrium, creatinine, CRP, AST, bilirubin, alkaline phosphatase, TSH, p-ionized calcium, PTH, Ca ++, and 25-OH vitamin D.
Side effects | Measured every four weeks through the study (for 5 months)
  Measuring a lot of posssible side effects to training and testosterone
Safety parameters - blood sample - testosterone level | Measured every four weeks through the study (for 5 months)
  Measuring levels of testosterone and safely parameter
Safety parameters - blood sample - hemoglobin level | Measured every four weeks through the study (for 5 months)
  Measuring levels hemoglobin
Safety parameters - blood sample - hematocrit level | Measured every four weeks through the study (for 5 months)
  Measuring levels of hematocrit
Safety parameters - blood sample - lipid profile | Measured every four weeks through the study (for 5 months)
  Measuring levels cholesterol
Safety parameters - blood sample - Potassium | Measured every four weeks through the study (for 5 months)
  Measuring levels of potassium
Safety parameters - blood sample - Natrium | Measured every four weeks through the study (for 5 months)
  Measuring levels of natrium
Safety parameters - blood sample - creatinine | Measured every four weeks through the study (for 5 months)
  Measuring levels of creatinine
Safety parameters - blood sample - CRP | Measured every four weeks through the study (for 5 months)
  Measuring levels of CRP
Safety parameters - blood sample - Aspartate aminotransferase (AST) | Measured every four weeks through the study (for 5 months)
  Measuring levels of aspartate aminotransferase (AST)
Safety parameters - blood sample - bilirubin | Measured every four weeks through the study (for 5 months)
  Measuring levels of bilirubin
Safety parameters - blood sample - alkaline phosphatase | Measured every four weeks through the study (for 5 months)
  Measuring levels of alkaline phosphatase
Safety parameters - blood sample - Thyreoid Stimulating Hormone (TSH) | Measured every four weeks through the study (for 5 months)
  Measuring levels of TSH
Safety parameters - blood sample - p-ionized calcium | Measured every four weeks through the study (for 5 months)
  Measuring levels of p-ionized calcium
Safety parameters - blood sample - PTH | Measured every four weeks through the study (for 5 months)
  Measuring levels of PTH
Safety parameters - blood sample - Ca ++ | Measured every four weeks through the study (for 5 months)
  Measuring levels of Ca2+
Safety parameters - blood sample - 25-OH vitamin D. | Measured every four weeks through the study (for 5 months)
  Measuring levels of vitamin D

CONTACTS AND LOCATIONS:
Overall Officials: Karsten Overgaard, M.D., Study Director — Herlev Hospital, Neurological Department N108
Locations (2):
- Denmark (2):
  - Karsten Overgaard, Hellerup, Danmark
  - Medical Dept. O, Geriatric Section, Herlev

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rasmussen RS, Midttun M, Zerahn B, Pedersen M, Rashid A, Ostergren PB, Paulin TK, Podenphanth TW, Karlsson LK, Rosendahl E, Ragle AM, Vinther A, Overgaard K. Testosterone and resistance training improved physical performance and reduced fatigue in frail older men: 1 year follow-up of a randomized clinical trial. Aging Male. 2024 Dec;27(1):2403519. doi: 10.1080/13685538.2024.2403519. Epub 2024 Sep 17. PMID 39289825
- [Derived] Rasmussen R, Midttun M, Kolenda T, Ragle AM, Sorensen TW, Vinther A, Zerahn B, Pedersen M, Overgaard K. Therapist-Assisted Progressive Resistance Training, Protein Supplements, and Testosterone Injections in Frail Older Men with Testosterone Deficiency: Protocol for a Randomized Placebo-Controlled Trial. JMIR Res Protoc. 2018 Mar 2;7(3):e71. doi: 10.2196/resprot.8854. PMID 29500160
- See also: Therapist-Assisted Progressive Resistance Training, Protein Supplements, and Testosterone Injections in Frail Older Men with Testosterone Deficiency: Protocol for a Randomized Placebo-Controlled Trial — https://www.researchprotocols.org/2018/3/e71
- See also: Testosterone serum levels in elderly fall-prone men do not correlate with age or performance in the 30 seconds chair stand test — http://www.jgerontology-geriatrics.com/article/view/285